CLINICAL TRIAL: NCT03381144
Title: A Phase I, Randomised, Double-Blind, Placebo-Controlled, Single Centre, 3-Part, Study Designed to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of Single and Multiple Ascending Doses of GDC-0334 and the Effect of Food on the Pharmacokinetics of GDC-0334 in Healthy Adult Subjects
Brief Title: A Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of Single and Multiple Ascending Doses of GDC-0334 and the Effect of Food on the Pharmacokinetics of GDC-0334 in Healthy Adult Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Molecule development was terminated
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GB40223; 2017-003498-33 (EudraCT Number)
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — GDC-0334

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1: GDC-0334 (Experimental): Participants in up to 7 cohorts will receive single, ascending doses of GDC-0334 under fasting conditions.
  Interventions: Drug: GDC-0334
- Part 1: Placebo (Placebo Comparator): Participants in up to 7 cohorts will receive single doses of placebo under fasting conditions.
  Interventions: Drug: Placebo
- Part 2: GDC-0334 (Experimental): Participants in up to 3 cohorts will receive single doses of GDC-0334 under fasting or fed conditions.
  Interventions: Drug: GDC-0334
- Part 2: Placebo (Placebo Comparator): Participants in up to 3 cohorts will receive single doses of placebo under fasting or fed conditions.
  Interventions: Drug: Placebo
- Part 3: GDC-0334 (Experimental): Participants in up to 4 cohorts will receive multiple, ascending doses of GDC-0334 under fasting or fed conditions.
  Interventions: Drug: GDC-0334
- Part 3: Placebo (Placebo Comparator): Participants in up to 4 cohorts will receive multiple doses of placebo under fasting or fed conditions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GDC-0334 — Part 1: GDC-0334 given orally with dose escalation between cohorts, based on emerging safety and pharmacokinetic (PK) data. Parts 2 and 3: doses to be based on the safety, tolerability, and PK data generated in the study. The dosing duration in Part 3 is planned to be at least 14 days, but no longer than 28 days.
  Arms: Part 1: GDC-0334; Part 2: GDC-0334; Part 3: GDC-0334
Drug: Placebo — Participants will receive GDC-0334-matching placebo.
  Arms: Part 1: Placebo; Part 2: Placebo; Part 3: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single-center, three-part study designed to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamic effects of single and multiple ascending doses of GDC-0334 and the effect of food on the pharmacokinetics of GDC-0334 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females. Females may be of non-childbearing potential or childbearing potential. Healthy females of childbearing potential must agree to use a highly effective method of contraception.
* Healthy males must agree to use an adequate method of contraception
* Body mass index of 18.0 to 32.0 kilograms per meter squared (kg/m^2) or, if outside the range, considered not clinically significant by the investigator
* Must be willing and able to communicate and participate in the whole study

Exclusion Criteria:

* Participants who have received any investigational medicinal product in a clinical research study within the previous 3 months
* Participants who are study site employees, or immediate family members of a study site or sponsor employee
* Participants who have previously been enrolled in this study. Participants who have enrolled in Part 1 are not permitted to enrol in Parts 2 or 3, and participants who have enrolled in Part 2 are not permitted to enroll in Part 3
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption >14 units per week (1 unit = ½ pint beer, 25 milliliters (mL) of 40% spirit or a 125-mL glass of wine)
* Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 6 parts per million (ppm) at screening or admission
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* Participants who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
* Clinically significant abnormal biochemistry, hematology or urinalysis as judged by the investigator
* Positive drugs-of-abuse test result at screening or admission
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus (HIV) results
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance of <70 milliliters per minute (mL/min) using the Cockcroft-Gault equation
* History of seizure
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, or psychiatric disorder, as judged by the investigator
* Participants with a history of cholecystectomy or gall stones (applies to any regimen where food effect is being explored)
* History of serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of active allergy requiring treatment, as judged by the investigator. History of hayfever is allowed unless it is active.
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Participants who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies in the 14 days or 5 half-lives, whichever is longer, before investigational medicinal product administration. Exceptions may apply on a case-by-case basis, if considered not to interfere with the objectives of the study, as agreed by the principal investigator and sponsor's medical monitor.
* History or presence of an abnormal electrocardiogram (ECG) that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third-degree heart block, or evidence of prior myocardial infarction, at screening or admission
* QT interval corrected using Fridericia's formula (QTcF) > 450 milliseconds (msec) demonstrated by at least two ECGs >30 minutes apart
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias such as structural heart disease, coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte abnormalities, or family history of sudden unexplained death or long QT syndrome
* Current treatment with medications that are well known to prolong the QT interval
* History of dermatographism
* Presence or history of clinically significant skin disorders, as judged by the investigator (Parts 1 and 3 only)
* History of trauma or surgery (laceration repair is not excluded) to the arm but not including wrist or hand injury/surgery (Parts 1 and 3 only)
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | From signing of informed consent until 30 days after the last dose of study drug (Up to approximately 42 days)
Severity of Adverse Events, as Graded per the World Health Organization (WHO) Toxicity Grading Scale | From signing of informed consent until 30 days after the last dose of study drug (Up to approximately 42 days)
Change from Baseline in Blood Pressure | Up to approximately 42 days
Change from Baseline in Heart Rate | Up to approximately 42 days
Incidence of Electrocardiogram (ECG) Abnormalities | Up to approximately 42 days
Incidence of Clinical Laboratory Abnormalities | Up to approximately 30 days
Incidence of Physical Examination Abnormalities | Up to approximately 42 days
Incidence of Neurological Examination Abnormalities | Up to approximately 31 days
Columbia-Suicide Severity Rating Scale (C-SSRS) - Part 3 Only | Up to approximately 42 days

SECONDARY OUTCOMES:
Elapsed Time from Dosing at Which GDC-0334 is First Quantifiable in a Concentration versus Time profile (Tlag ) | Up to approximately 35 days
Time to Maximum Plasma Concentration (Tmax) for GDC-0334 | Up to approximately 35 days
Maximum Observed Plasma Concentration (Cmax) for GDC-0334 | Up to approximately 35 days
Concentration at 24 hours Post-dose (C24) for GDC-0334 | Up to approximately 35 days
Concentration at 12 hours Post-dose (C12) for GDC-0334 | Up to approximately 35 days
Area Under the Plasma Concentration Curve from Time Zero to the Last Measurable Concentration (AUC0-t) for GDC-0334 | Up to approximately 35 days
Area Under the Plasma Concentration Curve from Time Zero Extrapolated to Infinity (AUC0-inf) for GDC-0334 | Up to approximately 35 days
Percentage of AUC0-inf Accounted for by Extrapolation to Infinity (AUC%extrap) for GDC-0334 | Up to approximately 35 days
Apparent Terminal Elimination Half-Life (t1/2) for GDC-0334 | Up to approximately 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Quotient Clinical Ltd, Clinical Research Unit, Nottingham, United Kingdom